CLINICAL TRIAL: NCT02161627
Title: Prospective, Multicenter, Randomized Double-blind Crossover Study Examining the Safety and Effectiveness of Spinal Cord Stimulation Incorporating Feedback to Treat Patients With Chronic Pain of the Trunk and/or Limbs in an Extended Trial
Brief Title: Safety and Effectiveness of Spinal Cord Stimulation With Automatic Control to Treat Chronic Pain in an Extended Trial
Acronym: Panorama
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBWSH1302; U1111-1157-5143 (Other: World Health Organization - Universal Trial Number)
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Pain
Keywords: spinal cord stimulation; automatic control
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automatic Control (Experimental): Automatic Control using Saluda Medical External Trial System
  Interventions: Device: Saluda Medical External Trial System
- Manual Control (Active Comparator): Manual Control using Saluda Medical External Trial System
  Interventions: Device: Saluda Medical External Trial System

INTERVENTIONS:
Device: Saluda Medical External Trial System
  Arms: Automatic Control
Device: Saluda Medical External Trial System
  Arms: Manual Control

SUMMARY:
The aims of the study are to compare automatic control of spinal cord stimulation with manual control in patients with chronic pain of the trunk and limbs

DETAILED DESCRIPTION:
Subjects will use the Saluda Medical External Trial System to compare automatic control of spinal cord stimulation with manual control in a randomized, blinded, crossover study.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in this study must meet the following inclusion criteria:

1. Have been diagnosed with chronic, intractable pain of the trunk and/or limbs (VAS ≥ 5), which has been refractory to conservative therapy for a minimum of 3 months.
2. Have been approved to undergo a trial of SCS.
3. Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician
4. Be on a stable dose (no new, discontinued, or changes in dose) of all prescribed pain medication for at least 4 weeks prior to the trial
5. Be 18 years of age or older at the time of enrollment
6. Be willing and capable of giving informed consent
7. Be willing and able to comply with study-related requirements, procedures, and visits
8. Females of childbearing age must have a negative urine pregnancy test at baseline

Exclusion Criteria:

Patients enrolled in this study must not meet the following exclusion criteria:

1. Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator
2. Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention and/or ability to evaluate treatment outcomes
3. Are not a surgical candidate due to a diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease or uncontrolled diabetes mellitus
4. Have a diagnosis of scoliosis that precludes lead placement
5. Have a condition, treatable with SCS, that requires leads to be inserted into the cervical region
6. Have an existing drug pump and/or SCS system or another active implantable device such as a pacemaker
7. Have a condition currently requiring or likely to require the use of MRI or diathermy
8. Have pain due to a malignant disease
9. Have a life expectancy of less than 1 year
10. Have an active systemic or local infection
11. Be allergic, or have shown hypersensitivity, to any materials of the neurostimulation system which come in contact with the body
12. Be pregnant or nursing (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile or be at least 2 years post-menopausal)
13. Have within 6 months of enrollment a significant untreated addiction to dependency producing medications or have been a substance abuser (including alcohol and/or illicit drugs)
14. Be concomitantly participating in another clinical study
15. Be involved in an injury claim under current litigation
16. Have a pending or approved worker's compensation claim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects With Improved Pain Relief and/or Stimulation Side Effects During the Automatic Control Arm Relative to the Manual Control Arm | 20 days
  After subjects experience both automatic and manual control after 20 days, subjects are asked to compare pain relief and stimulation side effects between the two arms of the study (blinded) in two separate domains using two 5-point Likert scales. The outcome measure for the primary objective is the percentage of subjects who report improved pain relief with no worsening of stimulation side-effects or improved stimulation side-effects with no loss of pain relief during the automatic control arm relative to the manual control arm. These subjects were considered successful for the primary outcome.

SECONDARY OUTCOMES:
Number of Adverse Events as a Measure of Safety | 20 days
Compare change from baseline of pain scores between automatic and manual control stimulation | 20 days
  Pain scores are obtained from the Visual Analog Scale (VAS) administered at baseline and after each arm of the study
Compare change from baseline of quality of life scores, between automatic and manual control stimulation | 20 days
  Quality of life scores are obtained from the Short Form - 36 (SF-36), and EuroQol-5D-5L questionnaires administered at baseline and after each arm of the study
Compare patient satisfaction with stimulation as measured on a 5-point Likert scale between automatic and manual control stimulation | 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Cousins, MD DSc, Principal Investigator — Pain Management Research Institute and Kolling Institute, University of Sydney at the Royal North Shore Hospital; Ashwini Sharan, MD, Principal Investigator — Department of Neurosurgery, Thomas Jefferson University Hospital
Locations (10):
- United States (10):
  - The Pain Center of Arizona, Phoenix, Arizona
  - Arizona Pain Specialists, Scottsdale, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Premier Pain Management, Shrewsbury, New Jersey
  - University Pain Management Center, Somerset, New Jersey
  - Center for Clinical Research, Winston-Salem, North Carolina
  - St Luke's Hospital, Neurosurgical Associates, Bethlehem, Pennsylvania
  - Performance Spine & Sports Physicians, East Norriton, Pennsylvania
  - Fox Chase Pain Management, Feasterville-Trevose, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania